CLINICAL TRIAL: NCT06850285
Title: Clinical Study on the Safety and Efficacy of Chimeric Antigen Receptor Gene Modified T Cells Targeting CD30 in the Treatment of CD30 Positive Relapsed/Refractory Lymphoma
Brief Title: CD30 CAR-T in the Treatment of CD30 Positive Relapsed/Refractory Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICT-CD30-2311-1
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma, B-Cell
Keywords: CD30 CAR-T; lymphoma;
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1 (Experimental): Subjects received a single low-dose CD30 CAR-T therapy(1*10^6/kg CAR+T cells)
  Interventions: Drug: chimeric antigen receptor gene modified T cells
- Group2 (Experimental): Subjects received a single low-dose CD30 CAR-T therapy(2*10^6/kg CAR+T cells)
  Interventions: Drug: chimeric antigen receptor gene modified T cells
- Group3 (Experimental): Subjects received a single low-dose CD30 CAR-T therapy(5*10^6/kg CAR+T cells)
  Interventions: Drug: chimeric antigen receptor gene modified T cells

INTERVENTIONS:
Drug: chimeric antigen receptor gene modified T cells — The rate of intravenous infusion of CD30 CAR T cells was 10 mL to 20 mL/min, and the infusion was performed using a blood transfusion apparatus with a filter screen. Use saline rinsing tube prior to infusion; Rinse the infusion bag with 10 mL~30 mL normal saline.
  Other Names: CAR-T

SUMMARY:
The is a prospective, open-label, dose-climbing clinical study assessing the efficacy and safety of CD30 CAR-T in the treatment of r/r CD30+ lymphoma. Plan to recruit 15 subjects with r/r CD30+ lymphoma。

DETAILED DESCRIPTION:
The goal of this clinical trial is to explore the effect of CD30 CAR-T on CD30 positive relapsed/refractory lymphoma. The main questions it aims to answer are:

To evaluate the safety of autologous CD30 CAR-T therapy in CD30-positive relapsed/refractory lymphoma; To evaluate the efficacy of autologous CD30 CAR-T therapy for CD30-positive relapsed/refractory lymphoma; To evaluate the metabolism of CD30 CAR-T cells in vivo; Preliminary evaluation of the correlation between CAR T cell dose and clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age≥15 years and ≤80years，female and male；
* CD30+ lymphocyte malignancies;
* CD30 expression >10% by immunohistochemistry；
* At least 1 measurable lesion can be measured according to theLugano 2014 evaluation criteria;
* Not suitable for autologous hematopoietic stem cell transplantation or recurrence after autologous hematopoietic stem cell transplantation;
* Not suitable for BV treatment or relapse after BV treatment, and the expression of CD30 was confirmed by histology;
* The estimated survival time ≥3 months;
* ECOG performance status 0-2，KPS>60%;
* Sufficient organ function：ALT，AST≤2.5×ULN，patients with liver invasion can be relaxed to ≤ 5 x ULN；serum total bilirubin<34 μmol/L；creatinine clearance rate>30 mL/min；EF≥40%；No pericardial effusion and obvious arrhythmia；SpO2≥92%；
* ALC ≥0.5×109/L，PLT>30×109/L，Hb>80 g/L and subjects had apheresis venous access and no contraindications for blood cell separation;
* MRI showed no central involvement of lymphoma;
* Patients with fertility must be willing to be able to use reliable contraceptive measures ;
* The subject or legal guardian can understand and voluntarily sign the written informed consent.

Exclusion Criteria:

* Lymphoma-associated hemophagic cell syndrome;
* Pregnant or lactating women, and women who have a pregnancy plan within six months;
* Hepatitis B（HBsAg、HBsAb、HBeAg、HBeAb、HBcAb），Hepatitis C（Anti-HCV），Anti-HIV Ⅰ/Ⅱ and anti-TP positive（Hepatitis B DNA test is negative except）;
* Suffered from other malignant tumors, except for for skin basal cell carcinoma, skin squamous cell carcinoma and cervical carcinoma in situ undergoing the radical treatment;
* Received Anti-CD30 Ab therapy within 4 weeks before enrollment;
* Unresolved > Grade 1 non-hematologic toxicity associated with any prior treatments;
* Active uncontrolled bleeding or a known bleeding diathesis;
* Autologous hematopoietic stem cell transplantation was performed within 6 weeks;
* Uncontrollable active bacterial or fungal infection；
* Known allergy to the study drug and its components;
* Suffer from active autoimmune diseases that require systemic treatment ;
* Persons with mental or mental illness who cannot cooperate with treatment and efficacy evaluation;
* Participated in other clinical studies within 1 months prior to this study;
* History of allogeneic hematopoietic stem cell transplantation;
* patients with any condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 months
  Including complete remission (CR) and partial remission (PR)
To evaluate safety and dose limiting toxicities (DLT) of autologous CD30 CAR-T and establish the recommended Phase dose | 28 days
  Incidence of DLTs and occurrence of study related adverse events

SECONDARY OUTCOMES:
Disease-free survival | 3years
  DFS was calculated from the first CAR-T cell infusion to death, progression of the disease, relapse or gene recurrence, whichever came first, or last visit.
Overall Survival | 3 years
  OS was calculated from the first CAR-T cell infusion to death or last follow-up

OTHER OUTCOMES:
The copy number of CD30 CAR-T cells | 12 months
  The copy number of CD30 CAR-T cells amplified in peripheral blood after administration

CONTACTS AND LOCATIONS:
Overall Officials: jia wei, Principal Investigator — Shanxi Bethune Hospital
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shangxi, China